CLINICAL TRIAL: NCT06316167
Title: Implementation of Mandatory Hiatoplasty in Sleeve Gastrectomy: Strategy for Gastro-Esophageal Reflux Disease (GERD) Risk Reduction
Brief Title: Mandatory Hiatoplasty in Sleeve Gastrectomy for Gastro-Esophageal Reflux Disease
Status: Recruiting | Type: Observational
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, GONZALEZ-OJEDA ALEJANDRO, Principal Investigator, Instituto Mexicano del Seguro Social
Other Study IDs: Hiatoplasty-2024
Record Dates: First submitted 2024-03-05; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Postgastrectomy Syndromes; Gastroesophageal Reflux
Keywords: Incidence; Complications; Bariatric surgery; Obesity
MeSH Terms: conditions — Postgastrectomy Syndromes; Gastroesophageal Reflux; Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about incidence of postoperative gastroesophageal reflux disease in mandatory hiatoplasty performed during gastric sleeve surgery.

The main question[s] it aims to answer are:

* Incidence of postoperative GERD in patients undergoing gastric sleeve with mandatory hiatoplasty
* Comparison of postoperative complication rates, including GERD

Participants will answer a follow-up questionnaire, about postoperative quality of life

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Gender indistinct.
* Overweight, obesity grade I, II, III, super obesity or super-super obesity.
* Underwent gastric sleeve with hiatoplasty for obesity management at a high volume Tijuana hospital dedicated to bariatric surgery.

Exclusion Criteria:

* Patient records with incomplete information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age of indistinct gender who underwent gastric sleeve with hiatoplasty for obesity or overweight management in a hospital center specialized in bariatric surgery in Tijuana, Baja California.
Sampling Method: Non-Probability Sample
Enrollment: 275 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants without postoperative GERD | 6 months
  To evaluate the efficacy of mandatory hiatoplasty performed during gastric sleeve surgery in reducing the incidence of postoperative gastroesophageal reflux disease (GERD) in patients undergoing this procedure in a hospital specializing in bariatric surgery in Tijuana, Baja California.

SECONDARY OUTCOMES:
Comorbidities in patients undergoing gastric sleeve with hiatoplasty | 6 months
  These patients usually have significant obesity, often accompanied by comorbidities such as type 2 diabetes, hypertension, sleep apnea, and gastroesophageal reflux disease (GERD).
Incidence of postoperative GERD in patients undergoing gastric sleeve with mandatory hiatoplasty | 6 months
  Hiatoplasty is often performed to reduce the risk of postoperative GERD by repairing a herniated hiatus during gastric sleeve surgery. However, the exact incidence of postoperative GERD can vary and depends on factors such as surgical technique, patient anatomy and postoperative management.
Comparison of postoperative complication rates, including GERD | 6 months
  Postoperative complications may include, but are not limited to, bleeding, infection, sleeve stenosis, and GERD recurrence. Comparison of complication rates between patients with and without mandatory hiatoplasty may provide insight into the effectiveness of this technique in mitigating specific risks.
Postoperative quality of life analysis | 6 months
  Questionnaire postoperative quality of life with the Bariatric Analysis and Reporting Outcome System (BAROS) Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: José Aldo Guzmán-Barba, MD, PhD, Study Chair — ALO Bariatrics. Gobernador Ibarra 9721, Zona Cacho, 22044, Tijuana, Baja California, México.; Alejandro López-Ortega, MD, PhD, Study Director — ALO Bariatrics. Gobernador Ibarra 9721, Zona Cacho, 22044, Tijuana, Baja California, México.; Helmut Heribert, MD, PhD, Principal Investigator — ALO Bariatrics. Gobernador Ibarra 9721, Zona Cacho, 22044, Tijuana, Baja California, México.; Isaac Esparza Estrada, MD, PhD, Study Chair — ALO Bariatrics. Gobernador Ibarra 9721, Zona Cacho, 22044, Tijuana, Baja California, México.; Sergio Jiram Vazquez-Sánchez, MD, Study Chair — Unidad de Investigación Biomédica 02, Unidad Médica de alta especialidad, Hospital de Especialidades Centro Médico Nacional de Occidente, Instituto Mexicano del Seguro Social, Guadalajara 44329, Mexico; Alejandro González-Ojeda, MD, PhD, Study Chair — Unidad de Investigación Biomédica 02, Unidad Médica de alta especialidad, Hospital de Especialidades Centro Médico Nacional de Occidente, Instituto Mexicano del Seguro Social, Guadalajara 44329, Mexico
Locations (1):
- Unidad de Investigación Biomédica 02, Unidad Médica de alta especialidad, Hospital de Especialidades Centro Médico Nacional de Occidente, Instituto Mexicano del Seguro Social, Guadalajara 44329, Mexico, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No
Data will be kept absolutely confidential

DOCUMENTS (1):
  • Study Protocol (2024-03-10): https://cdn.clinicaltrials.gov/large-docs/67/NCT06316167/Prot_000.pdf